CLINICAL TRIAL: NCT03649945
Title: An Open-label, Randomized Clinical Trial of Recombinant Human Endostatin (Endo) Combined With Chemotherapy Compared With Chemotherapy for Adjuvant Treatment of Esophageal Cancer
Brief Title: Endostatin Combined With Chemotherapy for Adjuvant Treatment of Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jie Ma, Director, First Affiliated Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRGX06
Record Dates: First submitted 2018-08-26; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Docetaxel; nedaplatin; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Group 1 (Active Comparator): Docetaxel plus Nedaplatin combined with Endostar
  Interventions: Drug: Docetaxel; Drug: Nedaplatin; Drug: Endostar
- Test Group 2 (Active Comparator): Docetaxel plus Nedaplatin
  Interventions: Drug: Docetaxel; Drug: Nedaplatin
- Control Group (No Intervention): No medicine intervention

INTERVENTIONS:
Drug: Docetaxel — 75mg/m2，3 weeks for one cycle，dosed on the first day of every cycle,totally 6 cycles
  Arms: Test Group 1; Test Group 2
Drug: Nedaplatin — 80 mg/m2,3 weeks for one cycle，dosed on the first day of every cycle,totally 6 cycles
  Arms: Test Group 1; Test Group 2
Drug: Endostar — 7.5mg/m2，once a day, continuously dosed for 14 days, then stop for 7 days,3 weeks for one cycle, totally 6 cycles
  Arms: Test Group 1

SUMMARY:
This is an open-label, randomized trial, it compares the efficacy and safety between apatinib combined chemotheray and chemotherapy for adjuvant treatment of esophageal cancer

ELIGIBILITY:
Inclusion Criteria:

* IIA-IIIC phase esophageal squamous cell carcinoma confirmed by histopathology and immunohistochemistry.
* R0 resection has been performed at least before 4 weeks.
* ECOG PS score: 0-1 points.
* Estimated survival time: at least 12 weeks.
* No radiotherapy, chemotherapy or molecular targeted therapy before.
* Main organs are functional, which meet the following criteria:

Blood Routine:

HB≥90 g/L（No blood transfusion within 14 days）, ANC≥1.5×109/L, PLT ≥80×109/L. Biochemical examination： ALB≥30g / L（No blood transfusion within 14 days）, ALT<2ULN； AST<2ULN TBIL≤1.5ULN； Plasma Cr≤1.5ULN；

* Volunteer with signed informed consent form, good compliance and good follow-up cooperation.
* Patients who the investigator believws they can benefit.

Exclusion Criteria:

* Those who have had other malignant tumors in the past or at the same time.
* Pregnant or lactating women.
* Patients with grade-II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTC interval ≥ 450 ms) and cardiac dysfunction according to NYHA criteria III to IV. Cardiac color Doppler examination: LVEF (left ventricular ejection) Score) <50%.
* Have clear gastrointestinal bleeding concerns (such as local active ulcer lesions, fecal occult blood ++), and a history of gastrointestinal bleeding within 6 months.
* Have a history of mental illness or psychotropic substance abuse.
* Patients who have participated in other drug clinical trials within 4 weeks.
* According to the investigator's judgment, patients who are at a risk or have accompanying disease.
* Patients who believe that they are unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
3 year disease-free survival rate | 3 years
  the percentage of the patients whose disease cannot be detected after curative therapy in three years

SECONDARY OUTCOMES:
overall survival | 3 years
  From the time of randomization to the time of death for any reason.

IPD SHARING:
Plan to Share IPD: Undecided